CLINICAL TRIAL: NCT07274709
Title: Emulation of the MONALEESA-2 Trial Using Specialty Oncology Electronic Health Records Databases
Status: Active, not recruiting | Type: Observational
Sponsor: Shirley Vichy Wang (Other)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Shirley Vichy Wang, Associate Professor, Brigham and Women's Hospital
Organization: Brigham and Women's Hospital (Other)
Other Study IDs: 2022P002556-ENC-MONALEESA-2; 75F40122C00181 (Other Grant/Funding Number: Food and Drug Administration)
Record Dates: First submitted 2025-11-20; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Advanced Breast Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Initiation of ribociclib plus letrozole: Exposure group
  Interventions: Drug: Initiation of ribociclib
- Initiation of letrozole: Reference group
  Interventions: Drug: Initiation of ribociclib; Drug: Initiation of letrozole

INTERVENTIONS:
Drug: Initiation of ribociclib — Initiation of ribociclib plus letrozole described in electronic health records is used as the exposure
Drug: Initiation of letrozole — Initiation of letrozole described in electronic health records is used as the reference
  Groups: Initiation of letrozole

SUMMARY:
Investigators are building an empirical evidence base for real world data through large-scale emulation of randomized controlled trials. The investigators' goal is to understand for what types of clinical questions real world data analyses can be conducted with confidence and how to implement such studies.

DETAILED DESCRIPTION:
Randomized controlled trials (RCTs) are generally regarded as the gold-standard of evidence for establishing efficacy of medical products. However, real-world data (RWD) are increasingly used to complement evidence from RCTs. Yet, to have confidence in the accuracy of non-interventional studies medical products and their outcomes in oncology, investigators need to know what questions can be validly answered, with which non-interventional study designs, and which analysis methods are appropriate, given the data that is available. Building on a process from the RCT DUPLICATE initiative1-4 EmulatioN of Comparative Oncology trials with Real-world Evidence (ENCORE) is part of the expansion project specific to oncology and aims to emulate 12 randomized oncology RCTs using multiple EHR data sources.

The purpose of this protocol is to describe the emulation of the MONALEESA-2 trial. MONALEESA-2 was a Phase III, double-blind, randomized study assessing the efficacy and safety of ribociclib (600 mg orally once daily on days 1-21 of a 28-day cycle, followed by 7 days off) in combination with letrozole (2.5 mg orally once daily, continuously) versus letrozole alone in postmenopausal women with hormone receptor-positive [estrogen receptor (ER) and/or progesterone receptor (PR)], human epidermal growth factor receptor 2-negative (HER2-) advanced breast cancer who had not received prior systemic treatment for their advanced disease.

ELIGIBILITY:
Study Period:

ENCORE database 1 (EDB1): Patient identification period: 01/01/2011-04/30/2024 with follow-up information through data cut-off date on 04/30/2024 ENCORE database 3 (EDB3): Follow-up information through June 2023 (there is no specific time period restrictions for patient eligibility) ENCORE database 4 (EDB4): Patient identification period: 10/01/2018-09/30/2023 with follow-up information through data cut-off date on 09/30/2023.

Inclusion Criteria:

* Age ≥18 years through 2017 to 2023
* Metastatic breast cancer
* Hormone receptor positive (ER/PR+)
* Untreated with systemic anticancer therapy for advanced disease
* ECOG performance status of 0 or 1
* HER2-negative

Exclusion Criteria:

* Prior treatment with CDK4/6 inhibitor
* Locally advanced (unresectable) or inflammatory breast cancer
* Non-breast cancer malignancy other than basal/squamous cell skin cancer or carcinoma in situ of cervix
* Prior adjuvant therapy for breast cancer
* Systemic anticancer therapy other than ribociclib or letrozole

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Postmenopausal women with hormone receptor (HR)-positive [estrogen receptor (ER) and/or progesterone receptor (PR)], human epidermal growth factor receptor 2 (HER2)-negative advanced breast cancer.
Sampling Method: Non-Probability Sample
Enrollment: 2495 (Estimated)
Dates: Start 2025-09-07 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Time to all-cause mortality/overall survival (OS) | From time of initiation of therapy through the earliest of death from any cause (the primary outcome of interest) or end of data availability (depending on specialty oncology registry data provider, end of data ranges from June 2023 to April 2024)
  Hazard ratio (95% CI)

CONTACTS AND LOCATIONS:
Overall Officials: Shirley Wang, PhD, ScM, Principal Investigator — Brigham and Women's Hospital; Denys Shay, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States